CLINICAL TRIAL: NCT06704659
Title: Study on Recurrent Breast Cancer and Repeated Radiation Therapy
Acronym: RAY-no-BAN
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Helsinki University Hospital, Finland (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1641/2024
Record Dates: First submitted 2024-11-21; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Recurrent Breast Carcinoma
Keywords: Breast cancer; Recurrence; Repeat radiation therapy; Radiation therapy
MeSH Terms: conditions — Breast Neoplasms; Recurrence | interventions — Radiotherapy; Mastectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Repeat breast conserving surgery and radiotherapy Arm (Experimental): The patients in this arm undergo repeat breast conserving surgery and partial breast radiotherapy
  Interventions: Radiation: Breast conserving surgey and radiotherapy
- Mastectomy Arm (Active Comparator): The patients in this arm undergo mastectomy
  Interventions: Procedure: Mastectomy

INTERVENTIONS:
Radiation: Breast conserving surgey and radiotherapy — The patients will undergo repeat Breast Conserving Surgery and Radiotherapy
  Arms: Repeat breast conserving surgery and radiotherapy Arm
Procedure: Mastectomy — The patients will undergo mastectomy
  Arms: Mastectomy Arm

SUMMARY:
This study explores whether recurrent breast cancer can be safely treated with breast-conserving surgery and repeated radiation therapy in cases where patients have previously undergone radiation. Traditionally, recurrent breast cancer has been treated by removing the entire breast. However, recent research has shown that in certain situations, it may be possible to preserve the breast.

The study will collect data on the safety of this treatment approach and its effects on patients. The treatment follows standard breast cancer care practices, involving 30 patients from Helsinki and Turku University Hospitals. Patients are carefully selected based on specific criteria, such as tumor size, localization, and prior treatment history. Special attention is given to the planning of radiation therapy and surgical techniques.

The goal is to develop new treatment strategies that allow breast preservation even in cases of recurrent breast cancer, providing patients with high-quality and individualized care.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a diagnosed breast cancer or tumor area in the breast with a maximum diameter of 3 cm, where a previous breast-conserving surgery has been performed (either invasive breast cancer or carcinoma in situ, DCIS).

The patient has only a local recurrence, and imaging studies show no suspicion of metastases outside the breast (preoperative staging N0M0).

At least 3 years have passed since the completion of prior radiation therapy. The new breast cancer can be technically treated with another breast-conserving surgery using a technique that does not require tissue transfer from areas opposite the removed tumor to restore the shape of the breast.

The patient is at least 55 years old at the time of surgery. The patient is willing to participate in the study. The patient is capable of providing informed consent.

Exclusion Criteria:

* A booster dose, also known as a "boost," was administered during prior radiation therapy.

Preoperative assessments suggest multifocal breast cancer, with the tumor area to be removed exceeding 3 cm.

The planned radiation therapy per the study protocol cannot be administered due to factors such as shoulder joint stiffness, a pacemaker located in the radiation field, or a skin condition (e.g., scleroderma).

The patient is unable to provide informed consent or is unwilling to participate in the study.

Metastases outside the breast (e.g., axillary or distant metastases) are present.

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
A treatment-limiting radiation therapy complication. | From the beginning of the radiotherapy until 30 days after finishing the therapy
  Any complication related to radiation therapy, that would limit completing the radiotherapy

SECONDARY OUTCOMES:
Quality of life | 5 years from surgery
  Patients are asked to complete a quality of life questionnaire before the surgery and at 3 months, 1 year, 3 years, and 5 years after the surgery
Second Breast Cancer Recurrence | 5 years from surgery
  The patients are surveilled for second breast cancer recurrence
Secondary malignancies | 5 years
  The patients are surveilled for any other secondary malignancy than breast cancer

CONTACTS AND LOCATIONS:
Locations (2):
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Turku University Hospital, Turku

IPD SHARING:
Plan to Share IPD: Undecided